CLINICAL TRIAL: NCT04697992
Title: Topical Tranexamic Acid Versus Topical Vitamin C With Microneedling in Periorbital Hyperpigmentation; Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Doaa Mohsen, Doaa Mohsen Fadl Morsy, Principal Investigator, teaching assistant at dermatology department, Kasr El Aini Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cosmo26
Record Dates: First submitted 2020-12-26; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Periorbital Hyperpigmentation
Keywords: Periorbital hyperpigmentation; Vitamin C; Tranexamic acid; Microneedling
MeSH Terms: interventions — Ascorbic Acid; Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: clinical trial, patients were divided into two groups, 30 each.
Who Masked: Outcomes Assessor
Masking Description: blinded investigators that assess grade of improvement at end of the study compared to baseline
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Experimental): one eye was treated with vitamin c 20% + microneedling a session was done every 2 weeks a total of 4 sessions (other eye was placebo treated with saline + microneedling).
  Interventions: Drug: vitamin c 20%
- group B (Experimental): one eye was treated with tranexamic acid 5 mg/ml + microneedling a session was done every 2 weeks a total of 4 sessions (other eye was placebo treated with saline + microneedling).
  Interventions: Drug: Tranexamic acid 5mg/ml

INTERVENTIONS:
Drug: vitamin c 20% — one eye was treated with vitamin c 20% + microneedling a session was done every 2 weeks a total of 4 sessions (other eye was placebo treated with saline + microneedling).
  Other Names: vitamin c 20% global cosmetic solutions
  Arms: group A
Drug: Tranexamic acid 5mg/ml — one eye was treated with tranexamin acid 5 mg/ml + microneedling a session was done every 2 weeks a total of 4 sessions (other eye was placebo treated with saline + microneedling)
  Other Names: kapron 500mg/ 5ml
  Arms: group B

SUMMARY:
Both vitamin C 20% and tranexamic acid 5mg/ml combined with microneedling were used for treatment of periorbital hyperpigmentation in a comparative pattern and both resulted in significant improvement of periorbital hyperpigmentation by dermoscopic and clinical evaluation with no statistically significant difference between them in addition to improvement of patients' visual analogue score (VAS) and dermatology life quality index (DLQI).

DETAILED DESCRIPTION:
Sixty patients with periorbital hyperpigmentation were enrolled, patients were divided into 2 groups; 30 each. clinical grading according to sheth et al.,2014 , dermoscopic evaluation, visual analogue score (VAS) and DLQI were done at week 0. Group A one side was treated with vit.c 20% + microneedling, other side saline+ microneedling (placebo). group B one side was treated with tranexamic acid 5mg/ml + microneedling, other side saline+ microneedling (placebo). A total of 4 sessions were done 2 weeks apart and follow up was one month after the last session (week 10) at which patient was evaluated using above mentioned parameters in addition to evaluation by 2 blinded investigators. At week 10 there was significant improvement of clinical grading and as evaluated by blinded investigators, VAS, DLQI, significant dermoscopic improvement in both vascular and pigmentary components of dark halos in sides treated with vit c and tranexamic acid compared to placebo but there was no statistically significant difference between both groups. The study concluded that tranexamic acid is a new safe effective modality in treatment of periorbital hyperpigmentation with results comparable to vitamin C.

ELIGIBILITY:
Inclusion Criteria:

* both genders.
* age ≥ 18 years.
* pigmentary, vascular and mixed types of dark halos

Exclusion Criteria:

* pregnancy and lactation
* patients who received treatment in the past 3 months
* patients with active dermatologic diseases or history of atopic dermatitis.
* history of allergy to tranexamic acid or vitamin c
* history of keloid or hypertrophic scars
* pure structural type of dark halos, pigmentary demarcation lines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
evaluation of effectiveness of tranexamic acid in periorbital hyperpigmentation | 10 weeks (patients are assissed 1 month after the last session)
  this is evaluated using dermoscopy (giving a score from 0 to 4, 0 = no improvement, 1=1-25% improvement, 2 =26- 50% improvement, 3=51-75% improvement, 4=>75% improvement)
evaluation of effectiveness of tranexamic acid in periorbital hyperpigmentation | 10 weeks (patients are assissed 1 month after the last session)
  clinical improvement by two blinded investigators (giving a score from 0 to 4, 0 = no improvement, 1=1-25% improvement, 2 =26- 50% improvement, 3=51-75% improvement, 4=>75% improvement)
evaluation of effectiveness of tranexamic acid in periorbital hyperpigmentation | 10 weeks (patients are assissed 1 month after the last session)
  clinical improvement by physician (grade from 0 to 4 according to sheth et al.,2014 where 0 no halos and 4 most severe)
evaluation of effectiveness of tranexamic acid in periorbital hyperpigmentation | 10 weeks (patients are assissed 1 month after the last session)
  dermatology life quality index (score from 0 to 30 the higher the worst)
evaluation of effectiveness of tranexamic acid in periorbital hyperpigmentation | 10 weeks (patients are assissed 1 month after the last session)
  patient visual analogue score (score from 0 to 10 the higher the worst)

CONTACTS AND LOCATIONS:
Locations (1):
- Doaa Mohsen, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No
im looking forward sharing the data but i have no plan yet